CLINICAL TRIAL: NCT06774820
Title: Self-locking Tenodesis of the Long Chief of the Biceps Vs. Lasso 360 Tenodesis in Arthroscopic Rotator Cuff Repair Rotator Cuff Repair
Acronym: BLAST1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Générale dAnnecy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-45-CGA
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Rotator Cuff Injury
Keywords: rotator cuff; biceps; long biceps tendon
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- self-blocking tenodesis (Experimental)
  Interventions: Procedure: self-blocking tenodesis
- arthroscopic tenodesis (Active Comparator)
  Interventions: Procedure: arthroscopic tenodesis

INTERVENTIONS:
Procedure: self-blocking tenodesis — the LHB tendon is detached from its origin in the superior labrum. This technique supports the self-locking mechanism of the LHB tendon in the bicipital groove by detaching the tendon from the Y-shaped superior glenoid, including the superior labrum. A radiographically visible suture will be attached to the proximal part of the LHB tendon to facilitate later localization of the LHB tendon during imaging (3-0 stainless steel, ethicon).
  Arms: self-blocking tenodesis
Procedure: arthroscopic tenodesis — LHB tendon is detached from its origin, and sutured. Next, the LHB tendon is fixed in the bicipital groove using a 360-lasso loop tenodesis technique. A radiographically visible suture will be attached to the proximal part of the LHB tendon to facilitate subsequent localization of the LHB tendon during imaging (3-0 stainless steel, ethicon).
  Arms: arthroscopic tenodesis

SUMMARY:
The aim of this study is to compare the clinical results and complications of self-locking biceps tenodesis and double 360 lasso loop biceps tenodesis for the treatment of long chief of biceps or superior labrum anterior-posterior (SLAP) tendon pathology during shoulder arthroscopy in patients undergoing arthroscopic rotator cuff repair. Currently, there is no consensus on the use of tenodesis versus tenotomy to treat pathology of the long head of the biceps during arthroscopic rotator cuff repair. Numerous studies have examined the clinical results of long biceps tenotomy versus long biceps tenodesis, and there is no evidence to date of superiority of either technique. At Clinique Générale, we use a new, innovative technique called autobloc tenodesis to treat pathologies of the long head of the biceps. There are no comparative studies between autobloc tenodesis of the biceps and biceps tenodesis. Given its potential advantages, self-locking biceps tenodesis could emerge as the new technique of choice for treating biceps longus tendon pathology, potentially reducing differences in outcomes such as Popeye deformity. The information provided by this study could potentially guide future clinical practice, helping surgeons to choose the most appropriate treatment for their patients suffering from long biceps tendon pathology.

ELIGIBILITY:
Inclusion Criteria:

* Full-thickness rotator cuff tear of the supraspinatus/infraspinatus tendon, diagnosed preoperatively by ultrasound, arthro-CT or MRI.
* Patients must be able to read and write in French in order to complete the questionnaires and sign the informed consent form.

Exclusion Criteria:

* Partial rotator cuff tear
* Massive and irreparable rotator cuff tear
* Grade 4 according to Goutallier classification of fatty degeneration of rotator cuff muscles
* Rupture of the long biceps
* Hourglass deformity of biceps tendon origin
* Osteoarthritis of the glenohumeral joint, defined by narrowing of the glenohumeral joint space or osteophytes, using AP radiography of the affected shoulder.
* Distance between acromion and humeral head measuring 6 mm or less, defined by Hamada classification as grade 2 or higher.
* Previous shoulder surgery.
* Dementia or inability to complete questionnaires and assessments.
* Pregnant, parturient or breast-feeding patients.
* Persons under legal protection (curatorship, guardianship, safeguard of justice).
* Persons deprived of their liberty by judicial or administrative measure
* Persons under psychiatric care
* Persons not affiliated to a social security scheme

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2027-11-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Constant score (CMS) | 1 year after surgery
  The CMS is a 100-point scale comprising four components, including a patient-reported section (pain 15 points and activity level 20 points), for a total of 35 points. Alongside this, there is a doctor-reported section (shoulder strength 25 points, range of motion 40 points) for a total of 65 points.

SECONDARY OUTCOMES:
American Shoulder and Elbow Surgeons Score | 3 months, 6 months, 1 year after surgery
  The ASES is a 100-point scale comprising 2 assessment dimensions: pain and activities of daily living.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Générale, Annecy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shirinskiy IJ, Boulidam D, Macken AA, van den Bekerom MPJ, Lafosse T, Buijze GA. Biceps lasso loop and self-locking tenodesis alongside repair of rotator cuff tears: randomised controlled trial study protocol (BLAST 1). BMJ Open. 2025 Nov 19;15(11):e106475. doi: 10.1136/bmjopen-2025-106475. PMID 41263857